CLINICAL TRIAL: NCT00738569
Title: A Pilot Study to Assess the Downregulation of HIV-1 Associated Chronic Inflammation in Patients With Limited Immunologic Responses When Raltegravir is Added to a Virologically Suppressed HAART Regimen
Brief Title: Assess the Downregulation of HIV-1 When Raltegravir is Added to a Virologically Suppressed HAART Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Merck HIV
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: HIV
Keywords: Chronic inflammation; memory cells; activated t-lymphocytes
MeSH Terms: interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raltegravir (Experimental)
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Raltegravir 400 mg PO BID for 12 months
  Other Names: Brand name is Isentress

SUMMARY:
The purpose of this study is to determine whether or not adding Raltegravir to a fully suppressive antiretroviral regimen will assist in reducing HIV-1 associated chronic inflammation and increase the t-lymphocyte memory cell pool.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. HIV-positive by Western blot or viral load
3. Viral load < 400 copies/ml
4. CD4+ T-lymphocyte count less than 350 cells/mm3 or change in CD4+ T-lymphocyte count < 100 cells/mm3 for at least one year on stable HAART with viral load < 400 copies/ml for the same period of time

Exclusion Criteria:

1. CD4+ T-lymphocyte count greater than or equal to 350 cells/mm3 or rise in CD4+ T-lymphocyte count greater than or equal to 100 cells/mm3 within one year of study entry
2. Viral load > 400 copies/ml
3. Allergy or resistance to raltegravir

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Quantitative changes in activated CD4+/CD8+ T-lymphocytes, pro-inflammatory cytokines and the central memory cell pool | 12 months

SECONDARY OUTCOMES:
Measure the change in circulating CD4+ and CD8+ T-lymphocytes | 12 months
Determine whether the circulating CD8+ T-lymphocyte count or the CD4+/CD8+ ratio can serve as a surrogate marker for suppression of chronic inflammation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Lichtenstein, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided